CLINICAL TRIAL: NCT02896296
Title: An Open-Label, Depot Buprenorphine (RBP-6000) Treatment Extension Study in Subjects With Opioid Use Disorder
Brief Title: Open-Label Treatment Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INDV-6000-301
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Opioid Use Disorder; Opioid-related Disorders
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- RBP-6000 (100/300 mg Flex) (Experimental): On Day 1 of the study all eligible subjects received a single subcutaneous (SC) injection of RBP-6000. Participants returned to the site for monthly injection visits every 28 days (-2/+7 days) for a total of up to 6 injections. Participants were not required to complete all 6 injections and could choose to terminate from the study at any time.
  For each injection, participants could receive either a dose of 100 mg RBP-6000 or 300 mg RBP-6000, based on the medical judgement of the investigator.
  Interventions: Drug: RBP-6000

INTERVENTIONS:
Drug: RBP-6000 — Monthly injections subcutaneously on alternate sides of participant's abdomen. Dose could be adjusted from 100 mg to 300 mg (or the reverse) based on the medical judgment of the investigator.
  Other Names: atrigel buprenorphine; extended-release buprenorphine

SUMMARY:
Study is to provide ongoing treatment with RBP-6000 and safety monitoring for subjects who complete the RB-US-13-0003 study (NCT02510014) and for whom a new treatment venue has not been identified or arranged.

DETAILED DESCRIPTION:
This is a multi-center, open-label, RBP-6000 treatment extension study in which subjects who have completed the End of Study (EOS) procedures for study RB-US-13-0003 are eligible. EOS assessments completed at the RB-US-13-0003 EOS visit serve as part of the screening visit for this study. In addition, subjects were requested to complete a Columbia Suicide Severity Rating Scale (C-SSRS) baseline/screening survey and a medical history and height was obtained.

The informed consent may be shared with subjects up to 2 months prior to the RB-US-13-0003 EOS visit, however should not be signed until all assessments for the EOS visit have been completed.

On Day 1, eligible subjects receive a subcutaneous (SC) injection of RBP-6000 at a low or high dose based on the medical judgment of the investigator. After the injection, vital signs and the injection site were assessed. Prior to departing the site, subjects were also assessed for adverse events (AEs) and use of concomitant medications (ConMeds).

Subjects return to the site for monthly injection visits every 28 days (-2 / +7 days) for a total of up to 6 injections (participants were not required to complete all 6 injections). At each subsequent visit (Injections 2 through 6) the following procedures / assessments were performed : urine pregnancy test performed for all female subjects who are of childbearing potential before each injection; previous injection site assessed for potential reaction and evidence of attempts to remove the depot; vital signs collected pre and post each injection; RBP-6000 injection, urine drug screen (UDS); C-SSRS since last visit assessment, counseling (manual-guided behavioral therapy); use of ConMeds; local injection site grading, subject self-assessment of injection site pain (Injection Site Pain Visual Analog Scale [VAS]), assessment for adverse events (AEs).

Laboratory tests (hematology, chemistry and urinalysis) may be requested by the Investigator on an ad-hoc basis in order to assess for AEs.

A subject's alternative treatment options were assessed at least two months before EOS at each visit.

At EOS or early termination (ET), the following assessments were performed: urine pregnancy test performed for all female subjects who are of childbearing potential; vital signs; previous injection site assessed for potential reaction and evidence of attempts to remove the depot; UDS; C-SSRS since last visit assessment, counseling (manual-guided behavioral therapy); use of ConMeds; assessment for AEs; a brief physical exam; height and body weight were measured and a subject's body mass index (BMI) and waist-to-hip ratio calculated; laboratory tests (hematology, chemistry, urinalysis).

Subjects were to be contacted by telephone approximately 4 weeks after EOS/ET for a safety follow-up assessment of AEs and use of ConMeds.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written consent to participate in this study.
2. Completed the End of Study Visit for the RB-US-13-0003 study (NCT02510014).
3. Be considered eligible in the medical judgment of the Investigator.
4. Females: Women of childbearing potential (defined as all women who are not surgically sterile or postmenopausal for at least 1 year prior to informed consent form (ICF)) must have a negative pregnancy test prior to enrollment and must agree to use a medically acceptable means of contraception from screening through at least 6 months after the last dose of investigational medicinal product (IMP).

   Males: Subjects with female partners of child-bearing potential must agree to use medically acceptable contraception after signing the ICF through at least 6 months after the last dose of IMP. Male subjects must also agree not to donate sperm during the study and for 6 months after receiving the last dose of IMP.
5. Subjects must agree not to take any buprenorphine products other than those administered during the current study throughout participation in the study.
6. Subjects must be willing to adhere to study procedures.

Exclusion Criteria:

1. Subject compliance issues during participation in the RB-US-13-0003 study which, in the opinion of the Investigator, could potentially compromise subject safety.
2. Women of childbearing potential who have a positive pregnancy test at RB-US-13-0003 at the end-of-study (EOS) visit, who are pregnant or breastfeeding, seeking pregnancy, or failing to use adequate contraceptive methods during the study.
3. History of suicidal ideation within 28 days prior to signing the ICF as evidenced by answering "yes' to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) "since last visit" assessment (completed in the EOS Visit for Study RB-US-13-0003), screening/baseline" assessment for the current study), or history of a suicide attempt (per the C-SSRS) in the 6 months prior to signing the ICF.
4. Taking any cytochrome P450 3A4 and 2C8 inducers and inhibitors, self-reported additional buprenorphine, or over the counter (OTC) and/or herbal supplements with the potential to prolong QTc within 28 days of Day 1 unless prior written approval was obtained from the Medical Monitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Director Clinical Development, Study Director — Indivior Inc.
Locations (29):
- United States (29):
  - Boyett Health Services, Hamilton, Alabama
  - Woodland International Research Group, Little Rock, Arkansas
  - Collaborative Neuroscience Network, Long Beach, California
  - Pacific Research Partners, Oakland, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Amit Vijapura, Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - Innovative Clinical Research, Lauderhill, Florida
  - Scientific Clinical Research, North Miami, Florida
  - Phoenix Medical Research, Prairie Village, Kansas
  - Louisiana Research Associates, New Orleans, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - Stanley Street Treatment and Resources, Fall River, Massachusetts
  - Adams Clinical Trials, Watertown, Massachusetts
  - Precise Research Centers, Inc., Flowood, Mississippi
  - St Louis Clinical Trials, St Louis, Missouri
  - Altea Research, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Neuro-behavioral Clinical Research, Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Rakesh Ranjan MD & Associates, Inc., Garfield Heights, Ohio
  - Pahl Pharmaceutical Professionals, Oklahoma City, Oklahoma
  - SP Research, PLLC, Oklahoma City, Oklahoma
  - CODA, Portland, Oregon
  - Keystone Clinical Solutions, Altoona, Pennsylvania
  - Carolina Clinical Trials, Charleston, South Carolina
  - Pillar Clinical Research, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rutrick D, Learned SM, Boyett B, Hassman D, Shinde S, Zhao Y. 18-Month efficacy and safety analysis of monthly subcutaneous buprenorphine injection for opioid use disorder: Integrated analysis of phase 3 studies. J Subst Use Addict Treat. 2023 Nov;154:209155. doi: 10.1016/j.josat.2023.209155. Epub 2023 Aug 30. PMID 37657559
- [Derived] Craft WH, Tegge AN, Keith DR, Shin H, Williams J, Athamneh LN, Stein JS, Chilcoat HD, Le Moigne A, DeVeaugh-Geiss A, Bickel WK. Recovery from opioid use disorder: A 4-year post-clinical trial outcomes study. Drug Alcohol Depend. 2022 May 1;234:109389. doi: 10.1016/j.drugalcdep.2022.109389. Epub 2022 Mar 9. PMID 35287034

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 208 subjects were screened across 25 sites, and of those, all 208 subjects entered the treatment period and received at least 1 dose of RBP-6000.
Period: Overall Study
Arm/Group | RBP-6000 (100/300 mg Flex)
Started | 208
Completed | 166
Not Completed | 42
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 19
Not completed — Pregnancy | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 10
Not completed — Site closing | 7
Not completed — Incarceration | 1
Not completed — Relocation | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Arm/Group | RBP-6000 (100/300 mg Flex)
Number analyzed (Participants) | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (11.47)
Age, Customized [Count of Participants; unit: Participants]
  >=18 and <30 years | 32
  >= 30 and < 45 years | 88
  >=45 and < 60 years | 71
  >= 60 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 198
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 78
  White | 129
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] — Population: Data missing for two participants
  cm
    number analyzed (Participants) | 206
    (all) | 173.26 (9.788)
Weight [Mean (Standard Deviation); unit: kg] | 78.41 (16.949)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Data missing for two participants
  kg/m^2
    number analyzed (Participants) | 206
    (all) | 26.12 (5.031)
Waist-to-Hip Ratio [Mean (Standard Deviation); unit: ratio] — Waist-to-hip ratio is the ratio of the waist circumference to hip circumference (calculated by dividing the waist circumference by the hip circumference). It is a measurement of abdominal fat distribution. Population: Records for one participant were missing baseline waist-to-hip ratio.
  ratio
    number analyzed (Participants) | 207
    (all) | 0.925 (0.0878)
Females of Childbearing Potential [Count of Participants; unit: Participants] — Population: Female participants only
  Participants
    number analyzed (Participants) | 70
    (all) | 40

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE) During the Treatment Period
Description: TEAE=any untoward medical occurrence that develops or worsens in severity after dispensation of the study drug and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= a marked limitation in activity. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 up to Week 29
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-6000 (100/300 mg Flex)
Number analyzed (Participants) | 208
Participants
  >=1 TEAE | 71
  >=1 TEAE related to study drug | 14
  >=1 serious TEAE | 5
  >=1 serious study treatment-related TEAE | 0
  Death | 0
  >=1 severe TEAE | 8
  TEAE leading to study treatment discontinuation | 1

2. Primary Outcome: Percentage Change From Baseline to Week 25 in Vital Signs
Description: Vital signs include:
  * systolic blood pressure (mmHg)
  * diastolic blood pressure (mmHg)
  * respiratory rate (breaths/minute)
  * pulse oximetry (%)
  * pulse rate (beats/min)
  * temperature (C)
Time Frame: Day 1, Week 25
Population: Safety analysis set. Participants with both baseline and Week 25 data are included.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | RBP-6000 (100/300 mg Flex)
Number analyzed (Participants) | 208
percentage change from baseline
  Systolic blood pressure: number analyzed (Participants) | 167
  Systolic blood pressure | 1.93 (11.208)
  Diastolic blood pressure: number analyzed (Participants) | 167
  Diastolic blood pressure | 2.61 (12.397)
  Pulse oximetry: number analyzed (Participants) | 167
  Pulse oximetry | 0.13 (1.377)
  Pulse rate: number analyzed (Participants) | 167
  Pulse rate | 6.04 (16.975)
  Respiratory rate: number analyzed (Participants) | 166
  Respiratory rate | 0.67 (8.360)
  Temperature: number analyzed (Participants) | 167
  Temperature | 0.02 (1.003)

3. Primary Outcome: Participants With Treatment-emergent Adverse Events (TEAEs) Pertaining to Laboratory Test Values
Description: TEAE=any untoward medical occurrence that develops or worsens in severity after dispensation of the study drug and does not necessarily have a causal relationship to the study drug. The number of participants with TEAEs specific to laboratory tests are summarized.
Time Frame: Day 1 up to Week 25
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-6000 (100/300 mg Flex)
Number analyzed (Participants) | 208
Participants
  Aspartate aminotransferase increased | 1
  Alanine aminotransferase increased | 1
  Blood cholesterol increased | 1
  Diabetes mellitus | 1
  Hepatic enzyme increased | 1
  Liver function test increased | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 29
Arm/Group | RBP-6000 (100/300 mg Flex)
All-Cause Mortality (participants affected / at risk) | 0/208
Serious Adverse Events (participants affected / at risk) | 5/208
Other Adverse Events (participants affected / at risk) | 0/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RBP-6000 (100/300 mg Flex) (N=208)
Pneumonia (Infections and infestations) | 3
Seizure (Nervous system disorders) | 1
Panic attack (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multi-center publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.

DOCUMENTS (2):
  • Study Protocol (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02896296/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT02896296/SAP_001.pdf